CLINICAL TRIAL: NCT05015062
Title: Effectiveness of a Mobile-based HIV Prevention Intervention for Rural and Low-income Population Involving Incentive Policy for Doctors in Liangshan, China: a Randomized Controlled Trial Protocol
Brief Title: Effectiveness of a Mobile-based HIV Prevention Intervention Involving Incentive Policy for Doctors in Liangshan, China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Yu Sun, Ph.D., Assistant Director, PKU China Center for Health Economic Research (CCHER), Peking University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 71833001
Record Dates: First submitted 2021-07-24; First posted 2021-08-20 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mobile-based intervention with standardized incentive (Experimental): Participants will receive biweekly messages containing HIV-related educational modules from village doctors who will receive standardized compensation for performing the work.
  Interventions: Behavioral: Mobile-based HIV-related educational message delivery
- Mobile-based intervention with performance-based incentive (Experimental): Participants will receive biweekly messages containing HIV-related educational modules from village doctors who will receive performance-based compensation for performing the work.
  Interventions: Behavioral: Mobile-based HIV-related educational message delivery; Behavioral: Incentive policies evaluation
- Control without intervention (No Intervention): Participants will not receive the mobile-based intervention

INTERVENTIONS:
Behavioral: Mobile-based HIV-related educational message delivery — HIV/AIDS awareness-raising and behavior-related cyclic messages will be delivered by the village doctors on a biweekly basis for 18 months.
  Arms: Mobile-based intervention with performance-based incentive; Mobile-based intervention with standardized incentive
Behavioral: Incentive policies evaluation — village doctors in Intervention A and B will receive different types of monetary compensation. Doctors in Intervention A will receive standardized compensation for completing their assigned tasks. Doctors in Intervention B will receive performance-based compensation whose amount depends on how well the participants perform on the follow-up questionnaires.
  Arms: Mobile-based intervention with performance-based incentive

SUMMARY:
This study will be carried out in Liangshan Yi Autonomous Prefecture, Sichuan province, China, using a single-blinded randomized controlled trial design to measure the effects of a mobile-based HIV-related information intervention on group HIV/AIDS prevention. Village doctors will be responsible for sending the HIV-related health education information to the participants. The aim of this study is to develop a generalizable, effective, acceptable, and convenient mobile-based information intervention model to improve HIV-related knowledge, attitudes, practices, and health outcomes in poverty-stricken areas in China and measure the impact of incentive policies on the work of village doctors in Liangshan, China.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older
* has mobile phone with internet service
* has and use WeChat and TikTok account regularly
* willing to provide informed consent
* speak Mandarin Chinese or Yi ethnic group's language

Exclusion Criteria:

* diagnosed with psychiatric disorders
* diagnosed with severe cognitive impairment
* diagnosed with severe physical disabilities
* has already attended or is currently attending another intervention program
* plan on moving out of Liangshan in the 18-month study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
HIV-related knowledge improvement | 18 months
  Result will be obtained by calculating weighted scores for the indicators in the HIV Knowledge Questionnaire 18 (HIV-KQ-18) to represent the participants' and their family members' level of knowledge measured by the baseline and follow-up questionnaires. The HIV-KQ-18 is a self-administered 18-item questionnaire; the possible scores range from 0 to 18, with 0-9 representing low HIV-related knowledge and 10-18 representing high HIV-related knowledge.
Comparison of the effectiveness of different financial compensations | 18 months
  The research team will compare the two interventions to determine what type of financial reward, standardized compensation or participant performance-based compensation, is more effective at incentivizing village doctors to deliver and promote the intervention content.

SECONDARY OUTCOMES:
Effectiveness of secondary knowledge transmission: HIV-related knowledge improvement of the participants' family members | 18 months
  The research team will examine the path of secondary knowledge transmission to the participants' family members by having the family members complete the HIV Knowledge Questionnaire 18 (HIV-KQ-18). The HIV-KQ-18 is a self-administered 18-item questionnaire; the possible scores range from 0 to 18, with 0-9 representing low HIV-related knowledge and 10-18 representing high HIV-related knowledge.
Behavioral changes: condom use | 18 months
  Assess the changes in participants' condom use via the Condoms Use Self-Efficacy Scale (CUSES), a 28-item self-reporting questionnaire using a 5-point scale scoring system in which 0 represents strongly disagree and 4 represents strongly agree.
Behavioral changes: substance use | 18 months
  Assess the severity, frequency and change of participants' substance use via the Drug and Abuse Screening Test (DAST), a 10-item questionnaire with scores range from 0 to 10; 0-2 representing low substance use and 9-10 representing severe substance use.
Health outcomes: HIV prevalence | 18 months
  Will be collecting regional data on HIV prevalence through collaboration with local departments.
Health outcomes: mental health | 18 months
  Assessed via the use of the Primary Care Evaluation of Mental Disorders (PRIME-MD) patient questionnaire, a self-reporting questionnaire consisting of 26 yes/no questions about the presence of various symptoms of different mental disorders.
Health outcomes: all-cause mortality | 18 months
  Will be collecting regional data on all-cause mortality through collaboration with local departments.
Social factors: quality of life | 18 months
  Measured via the use of EQ-5D-3L, a questionnaire comprised of 5 questions and a visual analogue scale to assess the participants' health-related quality of life. Each question has three possible answers corresponding to three levels of perceived problems. Level 1 indicates no problem and level 3 indicates extreme problems. The visual analogue scale is numbered from 0 to 100, with 0 representing "the worst health you can imagine" and 100 representing "the best health you can imagine"
Social factors: stigma towards HIV | 18 months
  Assessed via the use of the Internalized AIDS-Related Stigma Scale, a 6-item scale that offers a binary (yes/no) response to every item and the scores is computed as the sums of the items with 6 representing high stigmatization and 0 representing low stigmatization.
Social factors: perception of social support | 18 months
  Assess participants' social support in the community via the use of the Medical Outcomes Study Social Support Survey (MOS-SS), a self-reporting 19-item survey. The mean score of the 19 items will be calculated and transferred onto a 0-100 scale with higher scores indicating more support.
Retention of HIV-related knowledge | 18 months
  Measured by the HIV Knowledge Questionnaire 18 (HIV-KQ-18). The research team will ask all participants to complete the questionnaire every six months after the intervention period and compare their new scores with their previous score to examine their ability to recall information from the educational modules. The HIV-KQ-18 is a self-administered 18-item questionnaire; the possible scores range from 0 to 18, with 0-9 representing low HIV-related knowledge and 10-18 representing high HIV-related knowledge.
Feasibility: participants' use of social media applications | 18 months
  Feasibility of the intervention will be calculated by dividing the number of people who can use WeChat and TikTok by the total number of people living in the area.
Level of engagement | 18 months
  Measured by an original engagement and attendance scale. Participants will choose from a range 1 to 6, with 1 representing non-engaging and 6 representing highly engaging.
Study's acceptability and satisfaction | 18 months
  Assessed via an original 15-item questionnaire with rating scales (6 is Highly Satisfied and 1 is Highly Unsatisfied). Participants will be asked to rate and provide feedback on the intervention's content and method, including the effectiveness of the HIV-related knowledge modules, the time and method of information delivery, village doctors' attitude and competence, the design of the entire experimental intervention process, and more.
Cost-effectiveness of the intervention: | 18 months
  Data on the intervention's direct and indirect costs will be collected. Direct cost involves labor costs, research-related travel expenses, and village doctors' and participants' financial compensations. Indirect cost consists of the expenses on cell phone internet data. The date will then be used to evaluate the cost-effectiveness of both interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Guoen Liu, Principal Investigator — Peking University

REFERENCES:
- [Derived] Wang M, Liu G, Chen X, Ma S, Chen C. Effectiveness of a mobile-based HIV prevention intervention for the rural and low-income population involving incentive policy to doctors in Liangshan, China: a randomized controlled trial protocol. BMC Public Health. 2022 Sep 5;22(1):1682. doi: 10.1186/s12889-022-13930-2. PMID 36064390